CLINICAL TRIAL: NCT05647408
Title: Open Pilot Study to Evaluate the Bioavailability of Dexamethasone Administered Through Intranasal vs Intravenous Route.
Brief Title: Evaluation of the Bioavailability of Dexamethasone in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Edda Sciutto Conde, Principal Investigator, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BE20065-P
Record Dates: First submitted 2022-11-22; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Dexamethasone Administration; Intranasal Administration; Inflammation; Intravenous Drug Usage; Healthy Subjects
Keywords: dexamethasone; intranasal; pharmacokinetics; Bioavailability
MeSH Terms: conditions — Inflammation | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: 2 PERIODS, 2 TREATMENTS, 2 SEQUENCES, CROSSOVER 2X2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenously DMX (Active Comparator): Male and female volunteers received one dose of DXM. Drugs formulations employed were DXM phosphate injectable solution 8 mg/2 mL (Alin, Productos Farmaceuticos, Mexico). The drug was administered to 4 subjects intravenously (treatment A) according to a randomization list generated prior to the start of the clinical phase.
  Interventions: Drug: Dexamethasone
- Intranasally DMX (Active Comparator): Male and female volunteers received one dose of either DXM Drugs formulations employed were DXM phosphate injectable solution 8 mg/2 mL (Alin, Productos Farmaceuticos, Mexico). The drug was administered to 4 healthy subjects intranasally (treatment B). According to a randomization list generated prior to the start of the clinical phase.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — The nominal doses were similar, volunteers were randomly assigned to receive a single dose of DXM by IV bolus of 1.5 mL (equivalent to 6 mg of dexamethasone) or the same dose intranasally by using a Mucosal Atomization Device (MAD Nasal). allowing direct pharmacokinetic comparison without dose normalization. Venous blood samples were obtained via an indwelling catheter before administration and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12 and 24 h for DXM. Plasma was separated and frozen at -70 °C for further analysis.

SUMMARY:
The most important property of a dosage of a drug administration is its ability to deliver the active ingredient to the site of action in a quantity sufficient to exert the expected pharmacological effect. This ability is known as bioavailability. Dexamethasone is a drug with wide clinical use in patients with inflammatory pathologies (infectious or non-infectious). The main routes of administration are oral and intravenous. The intranasal route could be one more effective, less invasive that would allow to obtain a faster therapeutic concentration and in greater concentration in the lungs and in the central nervous system than the intravenous route, maintaining very similar systemic concentrations to those achieved intravenously. For these reasons, it is important to know the bioavailability of dexamethasone administered by this route in order to establish the best dosing regimen. The pilot study is of an exploratory nature (descriptive, comparative or informative), whose objective is to know the pharmacokinetic characteristics of a new route of administration of a drug in the study population to establish the pharmacokinetic parameters, and the comparison between the intranasal bioavailability against the intravenous administration by determining confidence intervals and calculating one-sided double t of Scuirmann.

Objetive: To evaluate the Absolute Bioavailability (for information purposes) of Dexamethasone 8 mg/2 ml Injectable Solution (Intranasal Route 6 mg/ 1.5 ml Vs Intravenous Route 6 mg/ 1.5 ml), according to the specific evaluation parameters and general under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible to participate in the study:

1. Age: 18 - 35 years (inclusive)
2. Health Status: Clinically healthy research subjects with the absence of clinically relevant abnormalities as identified by a medical history, physical examination, including determination of vital signs, a 12-lead electrocardiogram, and laboratory tests (which should be within normal values). allowed and corresponding validity, deviations will not be accepted)
3. Have not consumed any medication 2 days before starting hospitalization.
4. Signed and dated Informed Consent Form.
5. Body mass index of 18 -27 Kg/m2.
6. That it has been released from the COFEPRIS bioequivalence system database.
7. Signed non-pregnancy commitment letter (by female subjects)

Exclusion Criteria:

Subjects presenting any of the following circumstances will not be included in the study:

1. Clinical evidence or history of hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological disease or severe allergic reactions.
2. Any condition that may affect the absorption of the drug. (ex. Gastrectomy, Sprue, etc.)
3. Positive urine test for substances of abuse. Positive pregnancy test.
4. Use of products containing tobacco or nicotine 72 hours before and for the entire duration of the study.
5. Smoker (No more than 1 cigarette per day) or who has difficulty abstaining from tobacco consumption 72 hours before and for the entire duration of the study.
6. History of frequent excessive alcohol consumption 7 drinks per week for female subjects or 14 drinks per week for male subjects (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 4 months prior to the canvass.
7. Alcohol consumption before (48 hours) and during the study. (For this purpose, a breath test will be carried out with a breathalyzer prior to the start of each session).
8. Consumption of food or beverages that contain grapefruit and/or grapes or citrus fruits related to grapefruit (citrus) as well as carbonated foods or vegetarian diet or chocolate or coffee, from 3 days before the start of the study and until the last sample has been obtained.
9. Study drug treatment 30 days prior.
10. History of hypersensitivity to the study drug or its derivatives.
11. History of heparin sensitivity or heparin-induced thrombocytopenia.
12. A 12-lead resting EKG demonstrating a QTc of >450 msec at the time of screening. If the QTc exceeds 450 msec, the test should be repeated twice and the average of the three tests relative to the QTc should be used to determine subject eligibility (in the presence of clinical pathology findings).
13. Being participating in another study or having participated in another study without having elapsed at least the time equivalent to 7 half-lives of the drug administered in the previous study or without having elapsed 3 months. (whatever happens next)
14. Presence of use of prescription or non-prescription medications, dietary supplements, pre-study or herbal supplements, and hormonal methods of contraception (including oral, transdermal, injectable contraceptives, injectable progesterone, progestin implants). Women are expected to take appropriate precautions to prevent pregnancy and fetal exposure to a potentially toxic agent for the duration of the study (from the screening visit to the end of the study). Women of childbearing age will be informed that they must take the appropriate measures to prevent pregnancy during the study, such as the following: a) Willing to maintain abstinence (not having sexual intercourse) from 14 days before the start of the study to 28 days after the start of the study. end of study or b) Be willing to use two effective methods of birth control (condom, diaphragm, cervical cap, vaginal sponge, spermicides, non-hormonal IUD, tubal ligation, partner with vasectomy). Either of the two options from 14 days before the start of the study and up to 28 days after its conclusion. In no case may a lactating female subject participate.
15. Blood donation approximately 1 unit (500 mL) in a period of less than 90 days before the first study session.
16. Inability or refusal to comply with the indications described in this protocol.
17. Any other acute or chronic, medical or psychiatric, or laboratory condition that may increase the risk associated with the participation of the product to be administered or that may interfere with the interpretation of the study results and, in the Investigator's opinion, may compromise the participation of the subject in the study, including any type of recent hospitalization (1 month).
18. Results outside the normal values for the hematological, biochemical and laboratory tests carried out in the selection phase.
19. Subjects who have ingested a drug that induces or inhibits metabolism within the last two weeks prior to the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2021-11-06 (Actual); Study Completion 2021-11-13 (Actual)

PRIMARY OUTCOMES:
Absolute Bioavailability of Dexamethasone (6 mg/ 1.5 mL Intranasal Route vs. 6 mg/ 1.5 mL Intravenous Route) | 2 weeks
  The sample size used for this exploratory study (descriptive, comparative or informative) made it possible to determine the absolute bioavailability (with informative value), for which the bioavailability was compared in the 2 types of administration: Intranasal vs. Intravenous with a sample size of 8 research subjects, even though the ANADEVA is informative, the requirements regarding type I error (alpha), type II error (beta) and a minimum difference to detect between the 2 routes of administration: intranasal vs. IV.
  The realization of the present study allowed to know the pharmacokinetic and safety parameters of the drug Alin® administered by 2 different routes, as well as to determine the CVintra%.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Nacional Autonoma de Mexico, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No